CLINICAL TRIAL: NCT02776085
Title: Using Bedside Ultrasound to Measure the Optic Nerve Sheath Diameter in the Evaluation of Pediatric Patients With CSF Shunts
Brief Title: Bedside Ultrasound to Measure Optic Nerve Sheath Diameter in Pediatric CSF Shunts
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: ONSD
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2019-01

CONDITIONS: Cerebrospinal Fluid Shunts
Keywords: optic nerve sheath diameter; ultrasound; shunt failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Asymptomatic: Group of patients with CSF shunts who are evaluated for a reason other than concern for shunt failure. The optic nerve sheath diameter of these patients will be used as baseline measurements for children with CSF shunts.
- Symptomatic, Not Admitted: Group of patients with CSF shunts who are evaluated for concerns of shunt malfunction or failure, but either have shunt failure ruled out, or are felt to be safe for discharge to home. They are not admitted to the hospital. The optic nerve sheath diameter of these patients will be measured once in the emergency department.
- Symptomatic, Admitted: Group of patients with CSF shunts who are evaluated for concerns of shunt malfunction or failure, and then are admitted to the hospital secondary to these concerns. The optic nerve sheath diameter of these patients will be measured once in the emergency department or as close to admission as possible, and then measured again while they are still inpatient, but after they have an intervention performed (medical or surgical) to relieve their shunt malfunction or failure. These patients will have their initial optic nerve sheath diameters compared to the other two populations, but they will also have their initial and final optic nerve sheath diameters compared to each other.

SUMMARY:
Bedside ultrasound in the emergency department is useful for quick assessments of patients. One growing use is to measure the optic nerve sheath diameter of patients for whom increased pressure in the head is a concern. This study will look at the optic nerve sheath diameters of a specific population of pediatric patients with shunts that drain extra fluid from their heads.

DETAILED DESCRIPTION:
The particular interest of this study is the use of ultrasound to evaluate a child's optic nerve sheath diameter (ONSD), or the size of the covering around the nerve behind the eye. This covering expands when there is a higher than normal pressure inside the head. The group of interest on which this study focuses is the children with cerebrospinal shunts that drain extra fluid from their heads to other parts of the body (abdomen, heart, lungs) because the brain cannot drain all of the fluid like normal. When these shunts malfunction or fail, this can cause a backup of fluid in the brain, and raise the intracranial pressure (ICP) inside the skull. Depending on the degree of pressure buildup, this can be a surgical emergency due to pressure on the brain. Currently, computed tomography (CT) scans or magnetic resonance imaging (MRI) scans are used to diagnose the condition, but a quick screening tool, such as use of ultrasound to screen for elevated ICP in the emergency department, would be of great benefit to the patients to expedite care. Previous studies have explored the use of bedside ultrasound to evaluate the optic nerve sheath diameter in children with shunts. However, to date, there have been no reported prospective observational studies that compared before and after ultrasound measurements of the ONSD in patients in whom shunt failure is diagnosed and treated. Of note, this study is observational and the measurements taken with the ultrasound machine will not be used for clinical decision making. The measurements in this study will have no clinical impact on patient care. The use of ultrasound to measure the ONSD is an already accepted application of ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents, ages 6 months through 17 years who have a shunt and who present to the children's emergency department for evaluation and treatment.
* Children and adolescents, ages 6 months through 17 years who have a shunt and are directly admitted to the inpatient children's hospital from an outside facility.

Exclusion Criteria:

* Patients for whom the parents or guardians do not agree to participate in the study.
* Patients with any acute trauma to the eyes, face, or head.
* Severe anaphylactic allergy to ultrasound gel or Tegaderm

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients with cerebrospinal fluid shunts who are evaluated in the emergency department for any reason, or are admitted to the hospital through the neurosurgery clinic.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Compare the initial and final optic nerve sheath diameters measured by ultrasound in patients who are admitted for shunt failure | 3 days
  Patients will have their ONSD measured by ultrasound in the emergency department or immediately after admission. After they either receive antibiotics or shunt revision surgery, and are no longer symptomatic from shunt failure, their ONSD will be measured again and compared to the initial measurement.

SECONDARY OUTCOMES:
Compare the optic nerve sheath diameter measurements of asymptomatic patients vs symptomatic patients who are not diagnosed with shunt failure vs those are diagnosed with shunt failure and admitted. | 6 months
  The ONSD will be measured for all pediatric patients with CSF shunts who come to the emergency department, and then the average measurements of each group will be compared to the other two groups to evaluate if there are significant differences in the measurements.

OTHER OUTCOMES:
Physician Funduscopy Accuracy | 6 months
  The results of physician funduscopy of symptomatic patients will be compared to the imaging done for children to evaluate if physicians can visualize signs of increased intracranial pressure on funduscopic exam.

CONTACTS AND LOCATIONS:
Overall Officials: Christyn Magill, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No